CLINICAL TRIAL: NCT05761834
Title: Inflammation in Anderson-Fabry Disease and Hypertrophic Cardiomyopathy: A Comparative Study (FASHION STUDY)
Brief Title: FASHION Fabry Disease Hypertrophic Cardiomyopathy and Infammation
Acronym: FASHION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Liuzzo Giovanna, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4756
Record Dates: First submitted 2023-02-16; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Fabry Disease
Keywords: Hypertophic Cardiomyopathy
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Biospecimen Retention: Samples With DNA — to analyze plasma biomarkers, serum proteomic profile and transcriptomic analysis in peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Partecipants with Fabry Desease (FD): For each patient, at the time of enrollment, a blood sample will be collected and plasma levels of markers of inflammation, oxidative stress and cardiac remodeling will be determined (C-reactive protein, interleukin [IL]-6, IL-1β, IL-2, soluble vascular cell adhesion molecule, tumor necrosis factor [TNF], TNF receptor 1 and 2, Myeloperoxidase, calprotectin, uric acid, asymmetric dimethyl arginine, symmetric dimethyl arginine, matrix metalloprotease [MMP]-2, MMP-8 and MMP-9, galectin-1, galectin-3, B-type natriuretic peptide, midregional pro-atrial natriuretic peptide, monocyte chemoattractant protein-1).
  Serum proteomic analysis and transcriptomic analysis on peripheral blood mononuclear cells, investigating molecular mediators involved in inflammatory pathways will be also performed.
  Patients enrolled will also undergo a comprehensive 2D-echocardiography with Doppler, Tissue Doppler (TD) and speckle tracking analysis and 12-leads electrocardiogram.
  Interventions: Other: Sample blood and 2D-echocardiography with Doppler
- Partecipants with hypertrophic cardiomyopathy (HCM) systemic inflammation: For each patient, at the time of enrollment, a blood sample will be collected and plasma levels of markers of inflammation, oxidative stress and cardiac remodeling will be determined (C-reactive protein, interleukin [IL]-6, IL-1β, IL-2, soluble vascular cell adhesion molecule, tumor necrosis factor [TNF], TNF receptor 1 and 2, Myeloperoxidase, calprotectin, uric acid, asymmetric dimethyl arginine, symmetric dimethyl arginine, matrix metalloprotease [MMP]-2, MMP-8 and MMP-9, galectin-1, galectin-3, B-type natriuretic peptide, midregional pro-atrial natriuretic peptide, monocyte chemoattractant protein-1). Serum proteomic analysis and transcriptomic analysis on peripheral blood mononuclear cells, investigating molecular mediators involved in inflammatory pathways will be also performed.
  Patients enrolled will also undergo a comprehensive 2D-echocardiography with Doppler, Tissue Doppler (TD) and speckle tracking analysis and 12-leads electrocardiogram.
  Interventions: Other: Sample blood and 2D-echocardiography with Doppler

INTERVENTIONS:
Other: Sample blood and 2D-echocardiography with Doppler — Investigate whether patients with FD and HCM have a different inflammatory phenotype defined by plasma biomarkers, serum proteomic profile and transcriptomic analysis in peripheral blood mononuclear cells.
  Other Names: Tissue Doppler (TD) and speckle tracking analysis and 12-leads electrocardiogram.

SUMMARY:
In Fabry disease (FD) and hypertrophic cardiomyopathy (HCM) systemic inflammation recently gained attention as a possible key pathophysiologic process involved in the development of cardiac hypertrophy and progression of the disease. Differences in inflammatory profile between FD and HCM have never been investigated so far.

DETAILED DESCRIPTION:
This study investigate whether partecipants with FD and HCM have a different inflammatory phenotype defined by plasma biomarkers, serum proteomic profile and transcriptomic analysis in peripheral blood mononuclear cells. Moreover, the investigators sought to explore if a correlation exists between the inflammatory phenotype and the severity of cardiac phenotype cardiovascular events during 24 months of follow up.

This will be a prospective, multicenter, observational study. Adult partecipants with a genetically-proven diagnosis of FD and age-matched patients with a diagnosis of sarcomeric HCM will be enrolled, according to the following exclusion criteria:

1. Diagnosis Autoinflammatory disorders;
2. history of recurrent infections;
3. HIV infection;
4. Active cancer;
5. History of organ transplantation needing chronic immunosuppressor treatment. For each patient, at the time of enrollment, a blood sample will be collected and plasma levels of markers of inflammation, oxidative stress and cardiac remodeling will be determined (C-reactive protein, interleukin [IL]-6, IL-1β, IL-2, soluble vascular cell adhesion molecule, tumor necrosis factor [TNF], TNF receptor 1 and 2, Myeloperoxidase, calprotectin, uric acid, asymmetric dimethyl arginine, symmetric dimethyl arginine, matrix metalloprotease [MMP]-2, MMP-8 and MMP-9, galectin-1, galectin-3, B-type natriuretic peptide, midregional pro-atrial natriuretic peptide, monocyte chemoattractant protein.

Serum proteomic analysis and transcriptomic analysis on peripheral blood mononuclear cells, investigating molecular mediators involved in inflammatory pathways will be also performed. Partecipants enrolled will also undergo a comprehensive 2D-echocardiography with Doppler, Tissue Doppler (TD) and speckle tracking analysis and 12-leads electrocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Patients with confirmed genetic diagnosis of FD19;
* Patients with a known diagnosis of sarcomeric HCM adult (with pathogenic mutation in sarcomeric genes identified);
* Signed informed consent.

Exclusion Criteria:

* Age <18 years;
* Diagnosis of Autoinflammatory disorders;
* History of recurrent infections;
* HIV infection;
* Active cancer;
* History of organ transplantation needing chronic immunosuppressor treatment;
* Pregnancy
* Refusal to sign informed consent to study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with a genetically-proven diagnosis of FD and age-matched patients with a diagnosis of sarcomeric HCM will be enrolled.
  The spectrum of cardiomyopathies with hypertrophic phenotype encompasses heterogeneous diseases, including classic hypertrophic cardiomyopathy (HCM), due to sarcomere protein gene mutations, and several diseases mimicking HCM, such as Fabry cardiomyopathy.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-07-27 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Investigate the inflammatory phenotype of patients with FD and patients with HCM | 1 year
  Primary objective of the study is to investigate the inflammatory phenotype of patients with FD and patients with HCM.
  For each partecipants enrolled the investigators will record information about demographic and clinic data (age, gender, weight, height, hypertension, GLA gene mutation, sarcomeric genes mutation), conventional pharmacological therapy and specific therapy for FD patients such as Enzyme Replacement Therapy (α or β algasidase) or oral chaperon therapy (when it was started, therapeutic compliance).

SECONDARY OUTCOMES:
Correlation between the inflammatory phenotype and clinical, ECG and echocardiographic features, in both the diseases | 1 year
  Explore whether a correlation exists between the inflammatory phenotype and clinical, ECG and echocardiographic features, in both the diseases.
  Investigate the relationship between the inflammatory phenotype and the occurrence of MACEs (Major Adverse Cardiovascular Events, cardiovascular death, hospitalization for HF, new-onset atrial fibrillation, evolution to end-stage phase, sustained ventricular arrhythmias and/or bradyarrhythmias requiring pacemaker implantation, heart transplantation) during 24 months of follow-up in FD and HCM.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, Italy